CLINICAL TRIAL: NCT01259167
Title: JOBA & Chronic LOw BAck Pain
Brief Title: JOBA & Chronic LOw BAck Pain JOBA® & Chronic LOw BAck Pain JOBA® & Chronic LOw BAck Pain JOBA® & Chronic LOw BAck Pain
Acronym: JOBA-Loba
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Prof. Antonio Sgadari, Department of Gerontology, Geriatric and Physiatric Sciences, University Hospital "Agostino Gemelli"
Other Study IDs: 762/10
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-11

CONDITIONS: Low Back Pain
Keywords: JOBA, Low Back Pain, Physical Exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- BACK group: training with a traditional protocol of Therapeutic Physical Exercise
- Group "C".: Control group with sedentary people undergoing usual care.
- JOBA group: training with JOBA® Core Trainer

SUMMARY:
The purpose of this study was to assess whether a training program based on Joba® Core Trainer is effective in reducing pain and improving physical function and quality of life of subjects suffering from Chronic Low Back Pain.

DETAILED DESCRIPTION:
Background and rational

1. Definition Low back pain is a clinical condition characterized by pain felt between the bottom edge of the costal arch and the inferior gluteus folds, sometimes radiating to the back side of the thigh.

   It may be responsible for functional limitation and inability to perform normal activities of daily living. Low back pain is defined as acute if symptoms have a duration less than 4 weeks, sub-acute if the duration is between 4 weeks and 3 months, and chronic if it lasts beyond 3 months. It is considered recurrent when episodes shorter than 4 weeks alternate with periods of relief from pain.
2. Epidemiology Low Back Pain is the most common musculo-skeletal disorder, and, along with common cold, is the most frequent disease among humans.

   Up to 60-80% of population is expected to suffer from Low Back Pain at some time in life. Annual prevalence of Low Back Pain ranges from 30 to 50% amongst people in the working period of their life; out of these individuals, a percentage between 15 and 20% do necessitate medical assistance. Low Back Pain is the fifth-ranking cause of medical referral and the second symptomatic condition. A proportion ranging from 25 and 50% of patients with acute Low Back Pain will suffer from new pain episodes in the following year and 6-10% will progress toward a chronic form.Chronic Low Back Pain is responsible for about 75% of all medical expenses made for the treatment of all types of Low Back Pain. Direct annual costs (medications, medical visits, physiotherapy, hospitalizations) of Chronic Low Back Pain have been estimated to be approximately € 3.100 for patients (year 2002); indirect costs, mainly due to absence from work, represent about 85% of total costs and match up about € 17.600 for patient for year. In conclusion, Chronic Low Back Pain is a disease with very high prevalence and incidence, evenly affecting men and women in their 30's and 50's, which is extremely costly for individuals and society, both in terms of diagnostic interventions and treatments, and of reduction of productivity and functional limitation in everyday life.
3. Non-Pharmacologic treatments Non-Pharmacologic treatments of Chronic Low Back Pain include: acupuncture, back school, psychological interventions, functional restoration, interdisciplinary rehabilitation, interferential therapy, low-level laser therapy, lumbar support, massage, short wave diathermy, spinal manipulations, tractions, superficial heat, transcutaneous electrical nerve stimulations (TENS), ultrasound therapy, yoga and physical exercise.

   A recent meta-analysis based on 43 clinical controlled trials involving 3.907 subjects with Chronic Low Back Pain demonstrated that physical exercise is effective in reducing pain and improving functional level. The most recent Guidelines, published in October 20007, underline that, along with cognitive-behavioural therapy, spinal manipulations and interdisciplinary rehabilitation, physical exercise is the only non pharmacologic treatment having a positive effect on Chronic (or subacute) Low Back Pain.
4. Vertebral instability and physical exercise Several theories link the etiology of Low Back Pain clinical signs and symptoms to the mechanical instability of the lumbar spine. Stability of the lumbar spine requires both passive stiffness, through the osseous and ligamentous structures, and active stiffness, through "core" muscles, such as rectus abdominis, external oblique, internal oblique, transversus abdominis, quadratus lumborum, multifidi, psoas major, iliocostalis, gluteus major. It has been shown that therapeutic exercise improves vertebral stability through stretching and strengthening of "core" muscles, but also by enhancing neuromuscular proprioceptive facilitation. This is the reason why physical exercise programs usually do include strengthening and trunk-stabilizing exercises.
5. Joba® Core Trainer Joba® Core Trainer is a gym equipment which makes use of the counterbalance principle to efficiently engage trunk muscles, including both abdominals and trunk extensors. This equipment has been proved to be effective in improving cardio-respiratory fitness level, increasing resting energy expenditure, reducing weight and enhancing glycaemic control in diabetic patients. Furthermore it significantly strengthens diverse muscular groups (abdominals, trunk extensors, abductors, thigh flexors and extensors).

   Thus Core Trainer Joba® may represent a valuable alternative to traditional physical exercise protocols in the treatment of subjects with Chronic Low Back Pain
6. Study purpose The purpose of this study was to assess whether a training program based on Joba® Core Trainer is effective in reducing pain and improving physical function and quality of life of subjects suffering from Chronic Low Back Pain.
7. Materials and Methods 7a)Study design Randomized, one centre, single-blinded, clinical trial with three arms: JOBA group (training with JOBA® Core Trainer), BACK group (training with a traditional protocol of Therapeutic Physical Exercise) and Control group with sedentary people undergoing usual care (C).

7b)Subjects Subject attending the Physiatrist and Geriatric Outpatient Clinics of the Department of Gerontology, Geriatric and Physiatrist Sciences of the University Hospital "Agostino Gemelli" (Rome, Italy) with non-specific Low Back Pain, with or without sciatic irradiation, from at least 3 months. Exclusion criteria: functional or neurosensorial limitations which contraindicate or impede attending a physical exercise program (spondilolystesis higher than first degree, disk herniation more recent than 6 months, disk herniation for which surgical intervention is indicated, previous surgical intervention on spine, cognitive deterioration, terminal prognosis).

7c)Main outcome Perceived pain intensity. 7d)Secondary outcome

1. Quality of life
2. Level of physical function
3. Level of physical activity in everyday life
4. Neuro-muscular proprioceptive control of trunk-stabilizing muscles
5. Medication use/medical visits. 7e)Duration Twelve weeks.

8)Study phases 8a)Screening visit and enrolment Subjects to be enrolled into the study will be individuated during visits carried out at the Physiatrist and Geriatric Outpatient Clinics of the Department. Eligible subjects will be informed about the scope and methods of the study; those who will accept to participate will sign informed consent.

8b)Baseline assessment Patients will undergo a thorough medical visit (medical history, medication use, physical examination). The intensity of perceived low back pain, the level of physical functioning, and the quality of life will be measured (Mc Gill Pain Questionnaire-Short Form, Visual Analogue Scale, Roland-Morris Disability Questionnaire, Short-Form 36, respectively).The level of physical activity in everyday life (daily energy expenditure, physical activity >3 METs duration, active energy expenditure, average METs, number of steps, etc.) will be assessed by means of Metabolic Holter (Armband®) for a period of at least five consecutive days.Proprioceptive and neuro-muscular control of trunk muscles will be evaluated by means of a stabilometric, computerized table(Libra®).

8c)Randomization Subjects will be allocated to one of the three study groups according to a computerized randomization procedure with block of variable length.

8d)Intervention

1. JOBA Group: 3 sessions per week with JOBA® Core Trainer. Each session will last about 45 minutes (5-7 minute stretching exercises, 31' minutes with JOBA, 5-7 minute of stretching exercises). Speed of JOBA movements will progressively increase during the study period. All training session will take place in the Fitness Centre of the University Hospital "A. Gemelli".
2. BACK Group: 2 sessions per week (55 minutes each) of calistenic gymnastic with stretching, dynamic stabilization, and strengthening of trunk-stabilizing muscles, according to a standardized training protocol under the supervision of qualified technical personnel at the Fitness Centre.
3. Control Group (C): usual medical care according to the fore mentioned Outpatient Clinic standards.

8e)Intermediate assessment After 6 weeks, pain intensity, physical functioning, and quality of life will be re-evaluated; drug use and medical visits occurred from the baseline will be recorded.

8f)Final assessment After 12 weeks, subjects will undergo a complete medical visit and a new functional evaluation accordin to procedures already depicted for baseline (pain, physical function, quality of life, physical activity, proprioceptive control of the trunk, care-associated costs).

Blinding Due to the characteristics of the intervention, participants will be aware of the specific group the are allocated to (either traditional training or JOBA or usual care). However, baseline, intermediate, and final assessment will be carried out by a field researcher (a medicine doctor) uninformed of the allocation arm of the subject.

Sample size According to literature data it has been hypothesized that the intervention will produce a 20 (per cent) points increase in pain scale with respect to controls; using a probability of type I error of 5% (alfa=0.05, single-sided) and a power of 80% (beta=0.20), it can be estimated that each group should include 12 subjects (total sample size 12x3=36).

9)Analisi statistica Statistical analysis will be carried out on an intention-to-treat approach. Statistical analysis will be carried out using statistical software package SPSS/PC Vers. 18.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of low back pain (back pain, felt between the bottom edge of the costal arch and the inferior gluteus fold)
2. Chronic (with symptoms that persist for more than 12 weeks)
3. Not specific (i.e. not caused by specific pathophysiological mechanisms, such as infections, fractures, tumors, spinal canal stenosis)
4. With or without irradiation of the sciatic nerve

Exclusion Criteria:

1. Spondylolisthesis > First Instance
2. Osteoporosis with vertebral collapse
3. Herniated discs expelled for less than 6 months
4. Herniated discs with an indication for surgical treatment
5. Facet joint syndrome, high grade
6. Previous surgery to stabilize the spine in any section
7. Conditions that contraindicate the practice of physical exercise
8. Neuro-sensory limitations (blindness, deafness) that hinder the practice of physical exercise or communication (speech disorder)
9. Cognitive impairment
10. Diagnosis terminal
11. Change of residence over the next four months

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subject attending the Physiatrist and Geriatric Outpatient Clinics of the Department of Gerontology, Geriatric and Physiatrist Sciences of the University Hospital "Agostino Gemelli" (Rome, Italy) with non-specific Low Back Pain, with or without sciatic irradiation, from at least 3 months.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Fitness del Policlinico Agostino Gemelli di Roma, Roma, Italy